CLINICAL TRIAL: NCT00375817
Title: A Phase II, Open-Label, Randomized, Multicenter Study to Assess the Safety and Cardiovascular Effects of MyoCell Implantation by a Catheter Delivery System in Congestive Heart Failure Patients Post Myocardial Infarction(s)
Brief Title: Safety and Effects of Implanted (Autologous) Skeletal Myoblasts (MyoCell) Using an Injection Catheter = SEISMIC Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bioheart, Inc. (Industry)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: BMI-EU-02-008
Record Dates: First submitted 2006-09-11; First posted 2006-09-13 (Estimated); Last update posted 2007-10-12 (Estimated); Status verified 2007-10

CONDITIONS: Myocardial Infarction; Heart Failure, Congestive
MeSH Terms: conditions — Myocardial Infarction; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Myoblasts injection with MyoCath catheter

SUMMARY:
To assess the efficacy and safety of MyoCell therapy on myocardial function in congestive heart failure patients, post-myocardial infarction

ELIGIBILITY:
Inclusion Criteria:

* defined region of myocardial dysfunction related to previous MI (most recent MI at least 90 days prior to muscle biopsy involving the anterior, lateral, posterior or inferior walls, assessed by the presence of a Q-wave on the ECG & a large area of akinesia in the left ventricle, confirmed by either left ventricular angiography or echocardiography
* NYHA class II or III
* on optimal medical drug therapy for at least 2 months prior to study entry; defined by the most current ACC/AHA guidelines for the Evaluation & Management of chronic heart failure in the adult
* >=18 and <=75 years old
* need or feasibility for re-vascularization has been r/o by coronary or noninvasive stress testing within 30 days of screening, assessed using Dobutamine Stress Echocardiography
* able to undergo surgical biopsy of the skeletal muscle & successful culture of the harvested myoblasts
* well demarcated transmural myocardial scar (by echocardiography)Must have a minimum myocardial wall thickness of 5mm
* must have been fitted w/ an ICD in place for the duration of the study at least 6 months prior to muscle biopsy
* left ventricular EF at screening of >=20%, <=45% (by MUGA)
* willing & able to give written informed consent
* if female of childbearing potential, serum or urine pregnancy test must be negative w/in 2 weeks of study treatment

Exclusion Criteria:

* MI w/in 90 days of the muscle biopsy
* NYHA class I or IV
* CABG w/in 6 months (180 days) prior to scheduled MyoCell implantation
* PCI w/in 3 months (90 days) prior to scheduled MyoCell implantation
* aortic valve replacement
* heart failure secondary to valvular disease
* left ventricular mural thrombus
* known sensitivity to gentamicin sulfate and/or amphotericin-B
* previous experimental angiogenic therapy and/or myocardial laser therapy
* previous severe adverse reaction to nonionic radiocontrast agents
* exposure to any investigational drug or procedure w/in 1 month prior to study entry or enrolled in any concurrent study that may confound the results of this study
* serum creatinine >2.5 mg/dL or end stage renal disease
* active infectious disease and/or known to have tested positive for HIV, HTLV, HBV, HCV, CMV (IgM>IgG) and/or syphilis. If the panel includes antibodies to the HBV-cAg and HBV-sAg, then an expert will be consulted as to patient eligibility based on the patient's infectious status
* females who are pregnant or nursing or of childbearing potential who are unwilling to maintain contraceptive therapy for the duration of the study
* any illness which might affect patient's survival over the study follow up period or any illness which, in the investigator's judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of the study results
* patients on chronic immunosuppressive transplant therapy
* ICDs implanted less than 6 months prior to cellular implantation procedure. ICDs reprogrammed during the course of treatment and stable for less than 3 months. Patients fitted w/a Bi-V pacer are excluded.
* patients who, in the opinion of the investigator, are not suitable to participate, following review of the catheter information in appendix IV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Overall Objective
To assess the effect and safety of MyoCell™ therapy on myocardial function in congestive heart failure patients, post-myocardial infarction(s). Primary Safety Objective
The primary safety objective defined for this study is as follows:
The MyoCell™ implant will be considered safe if the number of serious adverse events at 3 months and 6 months is less than that seen in the control group (receiving standard medical therapy), and falling within levels set in the statistical analysis pla
Primary MyoCellTM Efficacy Objective
The primary efficacy objective of SEISMIC is to demonstrate the response to MyoCell™ implantation on the change in LVEF at 3 and 6 months by MUGA compared to baseline. Comparisons on LVEF will also be made between the two randomized groups (i.e. MyoCell

CONTACTS AND LOCATIONS:
Overall Officials: Jozef - Bartunek, MD, Principal Investigator — Cardiovascular Center, Aalst; Anthony - Gershlick, MD, Principal Investigator — Glenfield Hospital, University Hospitals of Leicester; Christoph - Hehrlein, MD, Principal Investigator — University of Freiburg; Carlos - Macaya, MD, Principal Investigator — Hospital Clinico San Carlos, Spain; Christoph - Nienaber, MD, Principal Investigator — University, Rostock, Germany; Nicholas - Peters, MD, Principal Investigator — St Mary's Hospital & Imperial College, London; Joachim - Schofer, MD, Principal Investigator — Universitaires Herzzentrum Hamburg, Germany; Patrick - Serruys, MD, Study Chair — Thorax Centre-Erasmus University, The Netherlands; Tomasz - Siminiak, MD, Principal Investigator — Cardiac & Rehabilitation Hospital at Kowanowko,Poland; Peter - Smits, MD, Principal Investigator — Medisch Centrum, Rijnmond Zuid, The Netherlands; J. - Waltenberger, MD, Principal Investigator — Academisch Ziekenhuis Maastrict, The Netherlands; Walter Van Mieghem, MD, Principal Investigator — ZOL Campus St. Jan, Genk, Belgium; Victor Legrand, MD, Principal Investigator — University Hospital, Liege, Belgium
Locations (1):
- Richard Spencer, Sunrise, Florida, United States